CLINICAL TRIAL: NCT04509895
Title: Minimally Invasive Calcaneal Fixation Via Sinus Tarsi Approach Vs Standard Lateral Extensile Approach in Calcaneal Fracture ( Randomized Controlled Trial )
Brief Title: Minimally Invasive Calcaneal Fracture Fixation vs Standard Lateral Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, peter mamdouh shehata, Resident doctor, Assiut University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: calcaneal fractures
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Calcaneus Fracture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lateral extensile approach in calcaneal fractures fixation (Experimental): Lateral extensile approach is the standard approach for intra-articular calcaneal fractures .
  Interventions: Procedure: Lateral extensile approach in calcaneal fractures fixation
- minimally invasive sinus tarsi approach in calc.fixation (Experimental): Sinus tarsi approach become one of the most frequently applied minimally invasive approaches.
  Interventions: Procedure: Minimally invasive sinus tarsi approach in calcaneal fractures fixation

INTERVENTIONS:
Procedure: Lateral extensile approach in calcaneal fractures fixation — The standard extended lateral approach with L-shaped incision was made in this group, which originated vertically from 5 cm over lateral malleolus or the midpoint between the fibula and Achilles tendon and ended on the base of the fifth metatarsal . The incision is made directly to the bone at the corner to create a full-thickness flap. Attention must be paid to protect the sural nerve and peroneal tendons as well.
  Arms: lateral extensile approach in calcaneal fractures fixation
Procedure: Minimally invasive sinus tarsi approach in calcaneal fractures fixation — An incision is made from the tip of the lateral malleolus toward the base of the fourth metatarsal bone. The incision lies in a plane between the superficial peroneal nerve and the sural nerve. Care is taken to bluntly dissect after the skin incision to protect the sural nerve or branches of the superficial peroneal nerve. By mobilizing the sinus tarsi fat pad dorsally, the incision was deepened. The extensor digitorum brevis muscle is sharply elevated off of the anterior process with the lateral root of the inferior extensor retinaculum and reflected dorsally and distally. The peroneus brevis and peroneus longus tendons are split, allowing exposure to the sinus tarsi and visualization of the posterior facet of the subtalar joint.
  Arms: minimally invasive sinus tarsi approach in calc.fixation

SUMMARY:
a comparison between the standard lateral extensile approach and minimally invasive sinus tarsi approach in this research.

DETAILED DESCRIPTION:
Calcaneal fracture occurred in about 2% of patients; they represented almost 60% of all tarsal fractures.

Calcaneal fractures are caused by high velocity Force to the heel, mostly vehicle accident or fall from height. There are many factors affect the fracture pattern: age of the patient, weight , type of fall . Male patients predominated (75%) and younger than 50 years. In most cases, these fractures are bilateral and conjoined with lumbar spine fractures.

According to the result of computed tomography (CT) scanning. The calcaneal fractures can be classified into 4 categories, among which the SANDERS TYPE Ⅱ and Ⅲ fractures are the most common types.2 Thus the development of effective and safe treatment strategies for these two fracture types has always been an issue among orthopedic surgeons.

The treatment of intra-articular calcaneal fractures has always been controversial. Currently open reduction and internal fixation through L-Shape extensile incision has been considered as the gold standard surgical therapy for calcaneal fractures. This approach provide a large view to expose the fracture, allowing accurate reduction of the deformed posterior facet and convenient placement of the plate to achieve stable fixation. Postoperatively, plaster cast is worn for 2 weeks, walking with the crutches for additional 8-12 weeks is prescribed, and return to work is achieved after 6-9 months. However, the high incidence (approximately 30%) of complications associated with this approach, including wound dehiscence and deep infection , remain a non-negligible problem .

To lower the wound complications , a minimally invasive approaches has been introduced such as percutaneously applied distraction systems K-wires or screw fixation of intra-articular fractures , the use of elizarov device , percutaneous arthroscopy assisted osteosynthesis and Sinus Tarsi approaches . The sinus tarsi approach has become one of the most frequently applied minimally invasive approaches because of its ability to provide adequate exposure for the posterior facet, the anterolateral fragment and the lateral wall. Wound complication rate with this approach have been reported to range from 0% to 15.4% . Nevertheless, the poor visualization of the lateral wall of the calcaneus through this small incision makes it difficult to insert the conventional plate for obtaining a stable fixation. Thus, the development of a plate that is adaptable to the anatomic characteristics of the calcaneus and sinus tarsi approach is important.

ELIGIBILITY:
Inclusion Criteria:

1. patients with calcaneal fractures according to Sanders classification, are Sanders type II or type III.
2. closed calcaneal fractures

Exclusion Criteria:

- 1)patients with calcaneal fractures classification according to sanders classification , are sanders type I or IV 2)patients who have systemic comorbidity as( cardic ,diabetec ,cirrhotic patients, etc.) or smokers or local lesion as (blisters,vasculopathy , swelling etc.).

3) open calcaneal fractures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
AOFAS( American association of foot and ankle score )for hind foot | baseline
  american association foot and ankle score

SECONDARY OUTCOMES:
Time needed before full weight bearing ( from 3 to 6 month ) | baseline
  the time the patient take for full weight bearing , usually take from 3 to 6 months in each arm
Radiological bohler angle | baseline
  restoration of bohler of hind foot
Wound complications | baseline
  wound dehiscence, infection, etc
Radiological gissane angle | Baseline
  Restoration of gissane angle of hind foot
Union rate | baseline
  the percentage of union in each arm

CONTACTS AND LOCATIONS:
Overall Officials: wael Y Eladly, professor, Study Chair — Assiut University
Locations (1):
- AssiutU, Asyut, Egypt

REFERENCES:
- [Result] Sanders R, Fortin P, DiPasquale T, Walling A. Operative treatment in 120 displaced intraarticular calcaneal fractures. Results using a prognostic computed tomography scan classification. Clin Orthop Relat Res. 1993 May;(290):87-95. PMID 8472475
- [Result] Cohen Z, Volpin G, Shtarker H. Surgical treatment of displaced calcaneal fractures Europian Instructional lectures, EFORT, 2011; 11: 199-214.
- [Result] Sanders RW, Clare MP. Fractures of the calcaneus in the Surgery of the Foot and Ankle, Coughlin MJ, Mann RA, Saltzman CL. (eds), Mosby Elsevier 8th ed. 2007; 2017-2073.
- [Result] Mitchell MJ, McKinley JC, Robinson CM. The epidemiology of calcaneal fractures. Foot (Edinb). 2009 Dec;19(4):197-200. doi: 10.1016/j.foot.2009.05.001. PMID 20307476
- [Result] Cao L, Weng W, Song S, Mao N, Li H, Cai Y, Zhou Q Jr, Su J. Surgical treatment of calcaneal fractures of Sanders type II and III by a minimally invasive technique using a locking plate. J Foot Ankle Surg. 2015 Jan-Feb;54(1):76-81. doi: 10.1053/j.jfas.2014.09.003. Epub 2014 Oct 18. PMID 25441282
- [Result] Backes M, Schepers T, Beerekamp MS, Luitse JS, Goslings JC, Schep NW. Wound infections following open reduction and internal fixation of calcaneal fractures with an extended lateral approach. Int Orthop. 2014 Apr;38(4):767-73. doi: 10.1007/s00264-013-2181-1. Epub 2013 Nov 27. PMID 24281853
- [Result] Yeo JH, Cho HJ, Lee KB. Comparison of two surgical approaches for displaced intra-articular calcaneal fractures: sinus tarsi versus extensile lateral approach. BMC Musculoskelet Disord. 2015 Mar 19;16:63. doi: 10.1186/s12891-015-0519-0. PMID 25886471
- [Result] Xia S, Lu Y, Wang H, Wu Z, Wang Z. Open reduction and internal fixation with conventional plate via L-shaped lateral approach versus internal fixation with percutaneous plate via a sinus tarsi approach for calcaneal fractures - a randomized controlled trial. Int J Surg. 2014;12(5):475-80. doi: 10.1016/j.ijsu.2014.03.001. Epub 2014 Mar 5. PMID 24607889
- [Result] Xia S, Wang X, Lu Y, Wang H, Wu Z, Wang Z. A minimally invasive sinus tarsi approach with percutaneous plate and screw fixation for intra-articular calcaneal fractures. Int J Surg. 2013;11(10):1087-91. doi: 10.1016/j.ijsu.2013.09.017. Epub 2013 Oct 5. PMID 24103451